CLINICAL TRIAL: NCT02540590
Title: Evaluation of Laser Speckle Contrast Imaging for Assessment of Oral Mucosal Blood Flow Following Periodontal Plastic Surgery: an Exploratory Observational Study
Brief Title: Post-operative Blood Flow Measurements of the Oral Mucosa
Acronym: LASCAM
Status: Completed | Type: Observational
Sponsor: Semmelweis University (Other)
Collaborators: Hungarian Scientific Research Fund (Unknown)
Responsible Party: Principal Investigator, Dr. Vag Janos, associate professor, Semmelweis University
Other Study IDs: 1/2013
Record Dates: First submitted 2015-08-25; First posted 2015-09-04 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Gingival Recession
Keywords: microcirculation; wound healing; tunnel technique; gingival recession; Mucograft; laser speckle contrast analyzer
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Mucograft: Laser speckle contrast imaging of the oral mucosa and wound fluid measurement before and after root coverage surgery. In this group the roots are covered by a combination of modified coronally advanced flap and xenograft collagen matrix (Mucograft).
  Interventions: Device: laser speckle contrast imaging of the oral mucosa; Device: wound fluid measurement
- CTG: Laser speckle contrast imaging of the oral mucosa and wound fluid measurement before and after root coverage surgery. In this group the roots are covered by a combination of modified coronally advanced flap and subepithelial connective tissue graft (CTG), which was harvested from the patient's palate.
  Interventions: Device: laser speckle contrast imaging of the oral mucosa; Device: wound fluid measurement

INTERVENTIONS:
Device: laser speckle contrast imaging of the oral mucosa — Non-invasive method to measure tissue blood perfusion applied for oral mucosa
  Other Names: LASCA, Perimed PSI
Device: wound fluid measurement — Wound fluid at the gingival sulcus was volumetrically measured by Periotron 8000 instrument using filter strip
  Other Names: Periotron

SUMMARY:
Our overall goal is to characterize the role of the microcirculation in healing oral mucosa after routinely applied surgery intervention in order to facilitate treatment. Using Laser Speckle Contrast Analysis (LASCA), which provides blood perfusion data, the investigators will have the possibility to detect functional alterations in gingival microcirculation in case of wound healing. After periodontal surgery, by means of the detection of microcirculation as a prognostic and diagnostic factor, the investigators can follow-up the healing procedure and obtain data so as to design e.g. the incision line that takes microvascular anatomy into account, thus result in better wound healing later on.

DETAILED DESCRIPTION:
In today's periodontal plastic surgery numerous flap designs with various grafting alternatives (auto-allo- or xeno-grafts) are routinely applied. In order to achieve uneventful primary intention healing and to allow for graft integration resulting in successful clinical outcomes it is important to apply optimized surgical techniques with suitable graft materials to address various clinical demands (e.g. recession coverage, enlargement of keratinized tissues, correction of periimplant soft tissue deficiencies). Graft exposure during soft- and hard tissue augmentation might occur before any chance of graft vascularization due to wound healing disturbances and lack of primary intention healing. The reasons of flap failure could be compromised flap circulation, which can be avoided by proper flap design, tension free flap advancement. The role of flap design on the gingival blood flow was investigated after surgery and found that the simplified papilla preservation flap resulted in faster recovery of the blood flow than the modified Widman flap surgery. In order to minimize trauma on surrounding tissues (i.e. flap) it is recommendable to use the least invasive method for flap preparation, which may also protect the underlining graft tissue and support quick vascularization. These guidelines led to develop a minimal invasive flap design for root coverage surgery, namely supraperiosteal envelope Tunnel technique, which was later modified by Azzi et al. to coronally advance the mucogingival complex in order to cover the inserted graft. Later it was further modified by introducing microsurgical approach. The question still remains to be answered how the Tunnelling technique can influence microcirculation of the healing gingiva and how the underlying graft tissue affects the overlying mucosal flap.

Recently a new non-invasive, two dimensional method, namely the laser speckle contrast analysis (LASCA) has been introduced to evaluate microcirculation of tissue. Clinical pilot studies are suggesting that this technique may be useful tool for assessing the proper circulation during surgical intervention and evaluating wound healing in the skin in human. This new method may let us monitor the entire surgical area real-time before and during the healing period.

ELIGIBILITY:
Inclusion Criteria:

* Having thin gingival biotype.
* Clinical diagnosis of multiple gingival recession
* Good general health

Exclusion Criteria:

* pregnancy,
* smoking,
* general diseases,
* take any antibiotics, antiinflammatory drugs, systemic steroids, biphosphonates, or any other medicines possibly influencing mucosal wound healing or any other products in the last three months (except contraceptives)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Caucasians subjects presenting multiple Miller Class I. and II. gingival recessions (Multiple Adjacent Recession Type Defects, MARTD) were recruited in the Department of Periodontology in Semmelweis University.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Postoperative blood flow changes of the oral mucosa | 6 months after surgery
  The blood flow changes were measured by Laser Speckle Contrast Analyzer (LASCA) before and after root coverage surgery (modified coronally advanced technique). The scale was an arbitrary unit (0-3000 LSPU) and the relative changes to the pre-operative measurement were calculated. Postoperative follow-up time-points were: 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 14, 17, 30, 60, 90, 120, 150, 180 days. The surgery was done with application of two different grafts (Mucograft-xenograft and connective tissue graft-autologous). The differences in postoperative blood flow changes were compared between the two graft-groups.

SECONDARY OUTCOMES:
Postoperative wound fluid changes of the oral mucosa | 6 months after surgery
  The wound fluid changes were measured by Periotron 8000 instrument. Using a filter strip to withdraw the fluid around the wound. The filter strip was then inserted into the Periotron machine to score the volume on the paper. The scores were in a range of 0-200 (arbitrary unit). Postoperative follow-up time-points were: 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 14, 17, 30, 60, 90, 120, 150, 180 days. The surgery was done with application of two different grafts (Mucograft-xenograft and connective tissue graft-autologous). The differences in postoperative wound fluid changes were compared between the two graft-groups.

CONTACTS AND LOCATIONS:
Overall Officials: Janos Vag, Principal Investigator — Semmelweis University, Dept. of Conservative Dentistry
Locations (1):
- Janos Vag, Budapest, Hungary